CLINICAL TRIAL: NCT01219283
Title: A Prospective Randomized Clinical Trial to Determine the Efficacy of 24 Chromosome Preimplantation Genetic Diagnosis
Brief Title: Study of the Efficacy of 24 Chromosome Preimplantation Genetic Diagnosis (PGD)
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RCT-2009-01
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Effect of PGD on Implantation Rates in IVF Cycles
Keywords: PGD; IVF

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from the male and female partners. Buccal swabs from infants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control (no PGD): Receive their planned IVF treatment without PGD. 2 morphologically best embryos are transferred.
- Case (PGD): Receive PGD in addition to their planned IVF Cycle. 2 morphologically best PGD normal embryos are transferred.

SUMMARY:
The purpose of this study is to determine if 24 chromosome preimplantation genetic diagnosis (PGD) increases implantation and delivery rates in couples attempting to conceive through in vitro fertilization (IVF).

DETAILED DESCRIPTION:
FISH based PGD techniques have provided little improvement in implantation and delivery rates. We believe that the use of 24 chromosome PGD, as compared to control (no PGD) will show a benefit to patients. This study is a randomized clinical trial that seeks to validate 24 chromosome PGD.

Patients that meet the eligibility criteria will be randomized prior to embryo transfer. In order to be randomized, the patient must have blastulated embryos suitable for biopsy on day 5. Half of the patients will received 24 chromosome PGD and will have 2 PGD normal embryos transferred. Half the the patients will receive no PGD and the 2 morphologically best embryos will be transferred. Follow up on pregnant patients will be a blood draw at approximately 9 weeks gestation and buccal swabs collected from the infant(s).

ELIGIBILITY:
Major Inclusion Criteria:

1. Age of female partner of < 43 years
2. Normal day-three FSH level (< 15 mIU/mL)
3. Normal uterine cavity
4. Sufficient ejaculated spermatozoa in male partner for ART
5. Maximum of one prior failed IVF cycle

Major Exclusion Criteria:

1. FSH level ≥ 15 mIU/mL
2. BMI greater than 32 kg/m2
3. Contraindication to gonadotropin stimulation
4. Unevaluated Ovarian mass
5. Need for surgical sperm removal
6. Any contraindication to undergoing in vitro fertilization
7. Age greater than 43 years
8. Presence of hydrosalpinges which communicate with the endometrial cavity
9. Clinical indication for PGD (undergoing IVF with PGD to rule out a known genetic defect)

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 500 patients attempting conception through IVF who have a maximum of one prior failed IVF cycle.
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Sustained Implantation Rate Per Embryo Transferred | Within 1 year
  Implantation rate per embryo transferred

SECONDARY OUTCOMES:
Clinical Pregnancy Rate and Delivery Rate per Treatment Cycle | Within 1 Year
  Clinical Pregnancy Rate and Delivery Rate per Treatment Cycle

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (3):
- United States (3):
  - Colorado Center for Reproductive Medicine, Lone Tree, Colorado
  - Reproductive Medicine Associates, Morristown, New Jersey
  - Reproductive Medicine Associates of PA at Lehigh Valley, Allentown, Pennsylvania

REFERENCES:
- [Derived] Scott RT Jr, Upham KM, Forman EJ, Hong KH, Scott KL, Taylor D, Tao X, Treff NR. Blastocyst biopsy with comprehensive chromosome screening and fresh embryo transfer significantly increases in vitro fertilization implantation and delivery rates: a randomized controlled trial. Fertil Steril. 2013 Sep;100(3):697-703. doi: 10.1016/j.fertnstert.2013.04.035. Epub 2013 Jun 1. PMID 23731996